CLINICAL TRIAL: NCT02622412
Title: Randomised Controlled Trial Testing the Effectiveness of a New Multi-professional Breathlessness sErvice for Patients With Any Advanced diSease Against Usual Care (BreathEase)
Brief Title: Evaluation of a Multi-professional Breathlessness Service for Patients With Breathlessness Due to Any Advanced Disease
Acronym: BreathEase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University Hospital Munich (Other); Helmholtz Zentrum München (Industry); University of Cambridge (Other); King's College London (Other)
Responsible Party: Principal Investigator, Claudia Bausewein, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01GY1331
Record Dates: First submitted 2015-10-31; First posted 2015-12-04 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Breathlessness; COPD; Cancer; Chronic Heart Failure; Interstitial Lung Disease
Keywords: Quality of Life; Palliative Therapy; Outpatient Services
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Neoplasms; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Patients randomised to the intervention group will get immediate access to the Multi-professional breathlessness service (MBS).
  Interventions: Other: Multi-professional breathlessness service (MBS)
- Control Group (Other): Patients randomised to the control group will get delayed MBS intervention. They will receive standard care and get access to the service after a waiting time of eight weeks.
  Interventions: Other: Delayed MBS Intervention

INTERVENTIONS:
Other: Multi-professional breathlessness service (MBS) — Patients visit the MBS twice. At week 1, delivered by palliative care specialists and respiratory disease specialists, patients receive an detailed assessment of breathlessness, relevant symptoms beyond breathlessness, psychosocial issues and carer burden. Recommendations are provided, and reviewed at the concluding visit in week 6 with palliative care specialists. In between these visits, weekly physiotherapy sessions focus on positioning, breathing techniques, exercise as well as pacing and fatigue management. Further support from the multi-professional expert team is given as needed.
  Arms: Intervention Group
Other: Delayed MBS Intervention — Patients will wait 8 weeks for start of intervention and will receive standard care in the meantime with access to respiratory medicine, general practitioners and palliative care services as needed. Standard care includes support by their general practitioners and disease orientated treatment (e.g. anti-obstructive treatment, oxygen supply if indicated, chemotherapy).
  Arms: Control Group

SUMMARY:
Breathlessness is a common and distressing symptom in patients with advanced diseases like cancer, chronic obstructive pulmonary disease (COPD), chronic heart failure (CHF) or lung fibrosis, which broadly impacts on patients' quality of life and may result in high burden for carers.

This single-blinded randomized controlled fast track trial evaluates the effectiveness of a multi-professional breathlessness service in patients with advanced and chronic diseases. The intervention group will get immediate access to the breathlessness service whereas the control group will receive standard care and get access to the service after a waiting time of eight weeks. Primary endpoints are mastery of breathlessness and quality of life, measured with the CRQ (Chronic Respiratory Questionnaire) as well as the reduction of symptom burden of patients and burden of carers. The evaluation of the cost effectiveness of the breathlessness service from the perspective of the German health system is a further study aim.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by breathlessness due to any advanced life-limiting and progressive disease, despite treatment of the underlying condition and
* Patients capable (in a cognitive and functional manner) to participate in the intervention including outpatient clinic and physiotherapist visits as well as self- management
* If patients are suffering from acute exacerbations of the underlying conditions, they are put on a waiting list for two to four weeks and are then entered into the trial.

Exclusion Criteria:

* Patients suffering from breathlessness due to chronic hyperventilation syndrome, asthma or any other unknown cause
* Cancer patients under concurrent initial or full dose systemic treatment or radiotherapy (except on maintenance therapy)
* Patients participating in any trial targeting the treatment of underlying conditions/ illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Mastery of breathlessness (CRQ mastery subscale) | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Change from baseline in Mastery of breathlessness (at week 8) measured with the Chronic Respiratory Disease Questionnaire (CRQ) in a face-to-face interview. Mastery represents one of the four CRQ domains containing 4 items. Patients rate their experience on each item a 7-point scale ranging from 1 (maximum impairment) to 7 (no impairment). The subscale "Mastery" is calculated by averaging the scores of the 4 items belonging to this subscale.
Quality of Life (CRQ) | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Change from baseline in Quality of Life (at week 8) measured with the CRQ. The CRQ contains 20 items across four domains: dyspnea, fatigue, emotional function, and mastery. Quality of life is calculated by adding all responses to all 20 items. Patients rate their experience on each item a 7-point scale ranging from 1 (maximum impairment) to 7 (no impairment)
Symptom Burden (IPOS) | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Change from baseline in palliative care needs and specific symptoms (at week 8) assessed with the Integrated Palliative Care Outcome Scale (IPOS). The IPOS includes 10 symptoms and 7 questions on patients and carers emotional situation, spiritual concerns, and provision of information and support. The overall profile score is the sum of the scores from each of the 17 questions.
Carers' burden of disease (ZBI) | From Baseline to End of Intervention (0, 8, 16 weeks)
  Change from baseline in carers' burden (at week 8) assessed with the Zarit Burden Inventory (ZBI), measuring personal strain and role strain. The revised version contains 22 items. Each item is a statement which the carer is asked to endorse using a 5-point scale. Response options range from 0 (never) to 4 (nearly always).

SECONDARY OUTCOMES:
Breathlessness severity (NRS) | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Change from baseline in breathlessness severity (at week 8) measured with numerical rating scales (NRS). The NRS will be used to assess breathlessness over the last 24 hours on average,at rest and on exercise. Responses on a rating scale range from 1 (no breathlessness) to 10 (strongest imaginable breathlessness).
Generic health-related quality of life (EQ-5D-5L) | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Change from baseline in patients' generic health-related quality of life measured with the EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The visual analogue scale of the EQ-5D-5L questionnaire ranges from 0 to 100 (with 0 representing the worst health the patient can imagine and 100 representing the best health the patient can imagine). Value sets of the EuroQol Group by time trade-off (TTO) will be used for scoring algorithm.
  The EQ-5D-5L is a standardized instrument applicable to a wide range of health conditions for use as a measure of health and is especially suited to cost effectiveness analyses.
Costs of health service utilization in Euros | From Baseline to Follow-Up (0, 8, 16, 28 weeks)
  Mean costs of intervention and control group (excluding study related costs) will be estimated. To calculate sum of costs in Euros per group to receive one aggregated outcome, firstly the following resource use data will be collected: Outpatient care, Medication, Medical aids, Inpatient care, Nursing home/hospice, Rehabilitation, Remedies (physiotherapy, massage, other), Formal care, Home help, Informal care, Work absenteeism, and early retirement. Secondly, resource use categories will be monetarily valued using unit cost and multiplied with the collected amount of resource use. Thirdly, mean costs in Euros per group will be calculated.
Patient survival measured in days | From randomization until death, up to end of study (24 months)
  Survival is defined as time from randomization to death irrespective of the cause of death. Participants who will not die during study course will be censored at the time of last contact which is planned for week 28 after last patient in. Survival status will be assessed by phone for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bausewein, Prof.Dr.med., Principal Investigator — Munich University Hospital
Locations (1):
- Hospital of the University of Munich, Department of Palliative Medicine, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Schunk M, Le L, Syunyaeva Z, Haberland B, Tanzler S, Mansmann U, Schwarzkopf L, Seidl H, Streitwieser S, Hofmann M, Muller T, Weiss T, Morawietz P, Rehfuess EA, Huber RM, Berger U, Bausewein C. Effectiveness of a specialised breathlessness service for patients with advanced disease in Germany: a pragmatic fast-track randomised controlled trial (BreathEase). Eur Respir J. 2021 Aug 26;58(2):2002139. doi: 10.1183/13993003.02139-2020. Print 2021 Aug. PMID 33509957
- See also: Study website — http://www.klinikum.uni-muenchen.de/Klinik-und-Poliklinik-fuer-Palliativmedizin/de/forschung/BreathEase/index.html
- See also: MBS website — http://www.klinikum.uni-muenchen.de/Klinik-und-Poliklinik-fuer-Palliativmedizin/de/klinik/Atemnot-Ambulanz/index.html